CLINICAL TRIAL: NCT02520713
Title: Multicenter Cohort Study To Evaluate Outcomes After Receipt of Targeted Therapy Matched to an Individualized Cancer Therapy (iCat) Recommendations in Children and Young Adults With Solid Tumors: The iCat2, GAIN Consortium Study
Brief Title: The iCat2, GAIN (Genomic Assessment Informs Novel Therapy) Consortium Study
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Katherine A. Janeway, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 15-169
Record Dates: First submitted 2015-06-18; First posted 2015-08-13 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Solid Tumor
Keywords: Pediatric Solid Tumor
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor and Germline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Genetic testing and GAIN report: All enrolled patients will submit specimens for sequencing and analysis.
  Interventions: Genetic: Genetic testing and GAIN report

INTERVENTIONS:
Genetic: Genetic testing and GAIN report — All patients enrolled will submit specimens for genetic analysis. If successful the report will be reviewed to look for possible recommendations and a GAIN report will be generated regardless of possible recommendations.

SUMMARY:
This research study is evaluating the use of specialized testing of solid tumors including sequencing. The process of performing these specialized tests is called tumor profiling. The tumor profiling may result in identifying changes in genes of the tumor that indicate that a particular therapy may have activity. This is called an individualized cancer therapy (iCat) recommendation. The results of the tumor profiling and, if applicable, the iCat recommendation will be returned.

DETAILED DESCRIPTION:
Patients with extra-cranial (not in the brain) solid tumors that are either difficult to diagnose or more difficult to treat are eligible to participate in this study. All enrolled patients will have targeted sequencing of tumor performed. Sequencing results will be reviewed for clinically significant findings including determination of whether any mutations exist that suggest potential for activity of a targeted therapy (iCat recommendation). Results will be returned to the patient's oncologist and follow-up data will be collected.

In this prospective multi-center cohort study, the primary objective is to describe the outcomes of pediatric patients with advanced solid tumors according to whether or not they received of targeted therapy matched to an iCat recommendation. The primary clinical outcome of interest is the endpoint of overall survival (OS), with progression-free survival and response rate (RR) as key secondary clinical outcome measures. To address this hypothesis, 825 patients will enroll from an anticipated 11 participating institutions over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age -- Age ≤ 30 years at time of initial qualifying solid tumor diagnosis
* Diagnosis -- Histologic diagnosis of solid malignancy (excluding brain tumors and lymphoma) that meets at least one of the following criteria:

  * Refractory, defined as tumor progression after initiation of standard first line therapy without having achieved a prior partial or complete remission OR Biopsy proven residual disease at the completion of planned standard initial front-line therapy.
  * Recurrent, defined as tumor progression after achieving a prior partial or complete remission
  * Newly diagnosed high risk disease, defined as having an expected event free survival of < 50% at 2 years.
  * Lacks definitive diagnosis or classical genomic findings after histologic review and standard molecular testing (rare tumor group).
* Examples include (eligibility not limited to these examples):
* Histology typically associated with a fusion in which fusion is not detected.
* Ewing-like sarcoma
* Undifferentiated sarcoma
* Inflammatory myofibroblastic tumor without ALK fusion
* Infantile fibrosarcoma without NTRK fusion
* Specimen Samples

  * Sufficient tumor specimen available to meet the minimum requirements for profiling from diagnosis or progression / recurrence

    --- OR
  * Surgery / biopsy planned as part of clinical care that is anticipated to yield sufficient material to meet the minimum requirements for profiling; OR
  * Patient has already had molecular profiling and patient has not yet started matched targeted therapy based on the report .

Exclusion Criteria:

* No Therapy Planned

  -- Patients who have declined further anticancer therapy will be excluded.
* Performance Status

  -- Patients with Lansky (age < 16 years) or Karnofsky (age ≥16 years) score < 50 will be excluded.
* Life Expectancy -- Patients with anticipated life expectancy < 3 months will be excluded.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High-risk, relapsed and refractory solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 18 months
  In pediatric patients with recurrent or refractory solid tumors who undergo successful molecular profiling, a) to describe the overall survival of patients by treatment group (iCatM, iCatUM and UM); b) to identify demographic, clinical, and genomic factors associated with overall survival from the time of relapse/progression (OSr); and c)to store tumor material, derived cell lines / xenografts, and blood samples for general sample banking and potential future research.

SECONDARY OUTCOMES:
Identification of the patient, clinical, and medication access factors associated with a) having an iCat recommendation and b) with receipt of matched targeted therapy. | 2 Years
Determination of factors associated with response and progression-free survival time by treatment group for patients with recurrent/refractory disease and measurable/evaluable disease. | 2 Years
Description of the frequency and range of molecular alterations in pediatric solid tumors at diagnosis and at relapse including a comparison of potentially targetable variants in paired tumor samples obtained from relapse and at initial diagnosis. | 2 Years
Determination of whether participation in a genomics study provides psychological well-being and whether that is associated with level of genomic comprehension and with receipt of an iCat recommendation. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Janeway, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Utah Childrens Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There is not plan to share IPD from this study at this time.